CLINICAL TRIAL: NCT01736566
Title: The MedSeq Project Pilot Study: Integrating Whole Genome Sequencing Into the Practice of Clinical Medicine
Brief Title: A Pilot Project Exploring the Impact of Whole Genome Sequencing in Healthcare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Human Genome Research Institute (NHGRI) (NIH); Baylor College of Medicine (Other); Duke University (Other)
Responsible Party: Principal Investigator, Robert C. Green, MD, MPH, Principal Investigator, The MedSeq Project, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MedSeq™; U01HG006500 (NIH)
Record Dates: First submitted 2012-08-17; First posted 2012-11-29 (Estimated); Results first posted 2018-11-07 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Healthy Adults (Full Study and Extension Phase); Hypertrophic Cardiomyopathy or Dilated Cardiomyopathy
Keywords: Primary Care; Cardiology; Hypertrophic Cardiomyopathy; Dilated Cardiomyopathy; Whole Genome Sequencing
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Cardiomyopathy, Dilated | interventions — Whole Genome Sequencing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Family History + Whole Genome Sequencing (Experimental): Doctors and their patients receive a Genome Report and an Annotated Family History Report.
  Interventions: Other: Family History + Whole Genome Sequencing
- Family History Only (Active Comparator): Doctors and their patients receive an Annotated Family History Report only.
  Interventions: Other: Family History Only

INTERVENTIONS:
Other: Family History + Whole Genome Sequencing — Doctors and their patients receive a Genome Report and a Family History report.
  There are two sections of the Genome Report:
  1. The General Genome Report, which include highly penetrant disease mutations, carrier status for recessive disease, and pharmacogenetic associations.
  2. The Cardiac Risk Supplement, which contain genetic information found in the genome regarding cardiac diseases or a risk of cardiovascular diseases that can help with the care of the patient.
  Extension Phase: Experimental: Family History + Whole Genome Sequencing
  *In the main study participants are randomized to either the Experimental or Other Arm, in the Extension phase of the study all participants are in the Experimental Arm.
  Arms: Family History + Whole Genome Sequencing
Other: Family History Only — Doctors and their patients receive a Family History report.
  Arms: Family History Only

SUMMARY:
The MedSeq™ Project seeks to explore the impact of incorporating information from a patient's whole genome sequence into the practice of clinical medicine. In the extension phase of MedSeq we are attempting increase our participant diversity by increasing targeted enrollment of African/African American patient participants.

DETAILED DESCRIPTION:
Whole genome sequencing (WGS) and whole exome sequencing (WES) services are currently available to and are being utilized by physicians and their patients in both research and clinical settings. The widespread availability and use of WGS and WES in the practice of clinical medicine is imminent. In the very near future, sequencing of individual genomes will be inexpensive and ubiquitous, and patients will be looking to the medical establishment for interpretations, insight and advice to improve their health. Developing standards and procedures for the use of WGS information in clinical medicine is an urgent need, but there are numerous obstacles related to integrity and storage of WGS data, interpretation and responsible clinical integration. MedSeq™ seeks to develop a process to integrate WGS into clinical medicine and explore the impact of doing so.

We believe that WGS will be used in many ways, including two distinct and complementary situations. In generally healthy patients, physicians will use the results of WGS to derive insight into future health risks and inform prevention and surveillance efforts, a category we refer to as General Genomic Medicine. In patients presenting with a family history or symptoms of a disease, physicians will use the results of WGS to interrogate particular sets of genes known to be associated with the disease in question, a category we refer to as Disease-Specific Genomic Medicine.

Beginning in fall 2012, we will enroll 10 primary care physicians and 100 of their healthy middle-aged patients to evaluate the use of General Genomic Medicine, and 10 cardiologists and 100 of their patients presenting with hypertrophic cardiomyopathy (HCM) or dilated cardiomyopathy (DCM) to evaluate the use of Disease-Specific Genomic Medicine. We will randomize physicians and their patients within each of the above models to receive clinically meaningful information derived from WGS versus current standard of care without the use of WGS.

MedSeq™ is comprised of three distinct but highly collaborative projects. Project 1 will enroll physicians and patients into the protocol, educate the physicians on basic genomic principles and safely monitor the use of genomic information in clinical practice. Project 2 will use a WGS analysis/interpretation pipeline to generate a genome report on each patient randomized to receive WGS in this protocol. Project 3 will examine preferences and motivations of physicians and patients enrolled, evaluate the flow and utilization of genomic information within the clinical interactions, and assess understanding, behavior, medical consequences and healthcare costs associated with the use of WGS in these models of medical practice.

In an extension phase of the study, we will 1) recruit approximately 10-15 patient-participants who self-identify as African or African American, whose physicians deem to be healthy. All will be placed in the whole genome-sequencing arm of the study. They will undergo the same activities as traditional MedSeq participants except for randomization. 2) We will conduct a targeted phenotype assessment on MedSeq Project patient-participants who are identified to have a monogenic finding. We plan to perform additional analysis by reviewing their medical records and looking specifically with their variant in mind to see if features associated with the variants were known prior to the study or were identified by further testing or by their physical during the course of the study.

This initiative will significantly accelerate the use of genomics in clinical medicine by creating and safely testing novel methods for integrating information from WGS into physicians' care of patients.

ELIGIBILITY:
Note for Age Eligibility:

* Cardiology patients 18 Years to 90 Years OR
* Primary Care Patients 40 Years to 65 Years (Adult, Senior)

Inclusion Criteria:

Primary Care

* Generally healthy (as defined by the primary care provider) adult patients at Brigham and Women's Hospital ages 40-65. All patients must be fluent in English.

Cardiology

* Patients in the Partners Healthcare System who are 18 years or older with a diagnosis of hypertrophic cardiomyopathy (HCM) or dilated cardiomyopathy (DCM) and a family history of HCM or DCM who previously had or who are candidates for targeted HCM or DCM genetic testing through routine clinical practice within Partners. All patients must be fluent in English.

Exclusion Criteria:

Primary Care

* Patients who do not meet the above criteria. Patients with cardiac disease or a progressive debilitating illness. Patients who are pregnant or patients whose spouses/significant others are pregnant. Patients with untreated clinical anxiety or depression (as measured by a Hospital Anxiety and Depression Scale (HADS) score > 11 administered at the baseline study visit.)

Cardiology

* Patients who do not meet the above criteria. Patients with a progressive debilitating illness. Patients who are pregnant or patients whose spouses/significant others are pregnant. Patients with untreated clinical anxiety or depression (as measured by a Hospital Anxiety and Depression Scale (HADS) score > 11 administered at the baseline study visit.)

Extension Phase - Additional Inclusion Criteria

Part 1:

* Above inclusion and exclusion criteria PLUS:
* Inclusion: Self-identify as African or African American.

Part 2:

Inclusion Criteria

* MedSeq participants determined to have a monogenic finding

Exclusion Criteria

* Participants not previously enrolled in MedSeq Project
* Participants not identified to have a monogenic finding

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2011-12 (Actual); Primary Completion 2016-11-04 (Actual); Study Completion 2021-01-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert C Green, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Biesecker LG. Opportunities and challenges for the integration of massively parallel genomic sequencing into clinical practice: lessons from the ClinSeq project. Genet Med. 2012 Apr;14(4):393-8. doi: 10.1038/gim.2011.78. Epub 2012 Feb 16. PMID 22344227
- [Background] Green ED, Guyer MS; National Human Genome Research Institute. Charting a course for genomic medicine from base pairs to bedside. Nature. 2011 Feb 10;470(7333):204-13. doi: 10.1038/nature09764. PMID 21307933
- [Background] Kohane IS, Masys DR, Altman RB. The incidentalome: a threat to genomic medicine. JAMA. 2006 Jul 12;296(2):212-5. doi: 10.1001/jama.296.2.212. No abstract available. PMID 16835427
- [Background] Khoury MJ, Berg A, Coates R, Evans J, Teutsch SM, Bradley LA. The evidence dilemma in genomic medicine. Health Aff (Millwood). 2008 Nov-Dec;27(6):1600-11. doi: 10.1377/hlthaff.27.6.1600. PMID 18997217
- [Background] Varmus H. Ten years on--the human genome and medicine. N Engl J Med. 2010 May 27;362(21):2028-9. doi: 10.1056/NEJMe0911933. No abstract available. PMID 20505183
- [Background] Evans JP, Meslin EM, Marteau TM, Caulfield T. Genomics. Deflating the genomic bubble. Science. 2011 Feb 18;331(6019):861-2. doi: 10.1126/science.1198039. No abstract available. PMID 21330519
- [Background] Hall MA, Camacho F, Lawlor JS, Depuy V, Sugarman J, Weinfurt K. Measuring trust in medical researchers. Med Care. 2006 Nov;44(11):1048-53. doi: 10.1097/01.mlr.0000228023.37087.cb. PMID 17063137
- [Background] Kaphingst KA, Facio FM, Cheng MR, Brooks S, Eidem H, Linn A, Biesecker BB, Biesecker LG. Effects of informed consent for individual genome sequencing on relevant knowledge. Clin Genet. 2012 Nov;82(5):408-15. doi: 10.1111/j.1399-0004.2012.01909.x. Epub 2012 Aug 7. PMID 22694298
- [Background] Carleton RN, Norton MA, Asmundson GJ. Fearing the unknown: a short version of the Intolerance of Uncertainty Scale. J Anxiety Disord. 2007;21(1):105-17. doi: 10.1016/j.janxdis.2006.03.014. Epub 2006 May 2. PMID 16647833
- [Background] Lipkus IM. Numeric, verbal, and visual formats of conveying health risks: suggested best practices and future recommendations. Med Decis Making. 2007 Sep-Oct;27(5):696-713. doi: 10.1177/0272989X07307271. Epub 2007 Sep 14. PMID 17873259
- [Background] Fagerlin A, Zikmund-Fisher BJ, Ubel PA, Jankovic A, Derry HA, Smith DM. Measuring numeracy without a math test: development of the Subjective Numeracy Scale. Med Decis Making. 2007 Sep-Oct;27(5):672-80. doi: 10.1177/0272989X07304449. Epub 2007 Jul 19. PMID 17641137
- [Background] Roter D, Larson S. The Roter interaction analysis system (RIAS): utility and flexibility for analysis of medical interactions. Patient Educ Couns. 2002 Apr;46(4):243-51. doi: 10.1016/s0738-3991(02)00012-5. PMID 11932123
- [Background] Brehaut JC, O'Connor AM, Wood TJ, Hack TF, Siminoff L, Gordon E, Feldman-Stewart D. Validation of a decision regret scale. Med Decis Making. 2003 Jul-Aug;23(4):281-92. doi: 10.1177/0272989X03256005. PMID 12926578
- [Background] Jarvik GP, Amendola LM, Berg JS, Brothers K, Clayton EW, Chung W, Evans BJ, Evans JP, Fullerton SM, Gallego CJ, Garrison NA, Gray SW, Holm IA, Kullo IJ, Lehmann LS, McCarty C, Prows CA, Rehm HL, Sharp RR, Salama J, Sanderson S, Van Driest SL, Williams MS, Wolf SM, Wolf WA; eMERGE Act-ROR Committee and CERC Committee; CSER Act-ROR Working Group; Burke W. Return of genomic results to research participants: the floor, the ceiling, and the choices in between. Am J Hum Genet. 2014 Jun 5;94(6):818-26. doi: 10.1016/j.ajhg.2014.04.009. Epub 2014 May 8. PMID 24814192
- [Background] Biesecker LG, Green RC. Diagnostic clinical genome and exome sequencing. N Engl J Med. 2014 Jun 19;370(25):2418-25. doi: 10.1056/NEJMra1312543. No abstract available. PMID 24941179
- [Background] Arndt AK, MacRae CA. Genetic testing in cardiovascular diseases. Curr Opin Cardiol. 2014 May;29(3):235-40. doi: 10.1097/HCO.0000000000000055. PMID 24717670
- [Background] Hwang KB, Lee IH, Park JH, Hambuch T, Choe Y, Kim M, Lee K, Song T, Neu MB, Gupta N, Kohane IS, Green RC, Kong SW. Reducing false-positive incidental findings with ensemble genotyping and logistic regression based variant filtering methods. Hum Mutat. 2014 Aug;35(8):936-44. doi: 10.1002/humu.22587. Epub 2014 Jun 24. PMID 24829188
- [Background] Lee IH, Lee K, Hsing M, Choe Y, Park JH, Kim SH, Bohn JM, Neu MB, Hwang KB, Green RC, Kohane IS, Kong SW. Prioritizing disease-linked variants, genes, and pathways with an interactive whole-genome analysis pipeline. Hum Mutat. 2014 May;35(5):537-47. doi: 10.1002/humu.22520. Epub 2014 Mar 6. PMID 24478219
- [Background] Vassy JL, Green RC, Lehmann LS. Genomic medicine in primary care: barriers and assets. Postgrad Med J. 2013 Nov;89(1057):615-6. doi: 10.1136/postgradmedj-2013-132093. No abstract available. PMID 24129030
- [Background] Berg JS, Amendola LM, Eng C, Van Allen E, Gray SW, Wagle N, Rehm HL, DeChene ET, Dulik MC, Hisama FM, Burke W, Spinner NB, Garraway L, Green RC, Plon S, Evans JP, Jarvik GP; Members of the CSER Actionability and Return of Results Working Group. Processes and preliminary outputs for identification of actionable genes as incidental findings in genomic sequence data in the Clinical Sequencing Exploratory Research Consortium. Genet Med. 2013 Nov;15(11):860-7. doi: 10.1038/gim.2013.133. Epub 2013 Oct 24. PMID 24195999
- [Background] Green RC, Berg JS, Grody WW, Kalia SS, Korf BR, Martin CL, McGuire AL, Nussbaum RL, O'Daniel JM, Ormond KE, Rehm HL, Watson MS, Williams MS, Biesecker LG; American College of Medical Genetics and Genomics. ACMG recommendations for reporting of incidental findings in clinical exome and genome sequencing. Genet Med. 2013 Jul;15(7):565-74. doi: 10.1038/gim.2013.73. Epub 2013 Jun 20. PMID 23788249
- [Background] McGuire AL, Joffe S, Koenig BA, Biesecker BB, McCullough LB, Blumenthal-Barby JS, Caulfield T, Terry SF, Green RC. Point-counterpoint. Ethics and genomic incidental findings. Science. 2013 May 31;340(6136):1047-8. doi: 10.1126/science.1240156. Epub 2013 May 16. No abstract available. PMID 23686340
- [Background] McGuire AL, McCullough LB, Evans JP. The indispensable role of professional judgment in genomic medicine. JAMA. 2013 Apr 10;309(14):1465-6. doi: 10.1001/jama.2013.1438. No abstract available. PMID 23571582
- [Background] Rehm HL. Disease-targeted sequencing: a cornerstone in the clinic. Nat Rev Genet. 2013 Apr;14(4):295-300. doi: 10.1038/nrg3463. Epub 2013 Mar 12. PMID 23478348
- [Background] Krier JB, Green RC. Management of incidental findings in clinical genomic sequencing. Curr Protoc Hum Genet. 2013;Chapter 9:Unit9.23. doi: 10.1002/0471142905.hg0923s77. PMID 23595601
- [Background] MacRae CA. Action and the actionability in exome variation. Circ Cardiovasc Genet. 2012 Dec;5(6):597-8. doi: 10.1161/CIRCGENETICS.112.965152. No abstract available. PMID 23250897
- [Background] Song T, Hwang KB, Hsing M, Lee K, Bohn J, Kong SW. gSearch: a fast and flexible general search tool for whole-genome sequencing. Bioinformatics. 2012 Aug 15;28(16):2176-7. doi: 10.1093/bioinformatics/bts358. Epub 2012 Jun 23. PMID 22730434
- [Background] Green RC, Berg JS, Berry GT, Biesecker LG, Dimmock DP, Evans JP, Grody WW, Hegde MR, Kalia S, Korf BR, Krantz I, McGuire AL, Miller DT, Murray MF, Nussbaum RL, Plon SE, Rehm HL, Jacob HJ. Exploring concordance and discordance for return of incidental findings from clinical sequencing. Genet Med. 2012 Apr;14(4):405-10. doi: 10.1038/gim.2012.21. Epub 2012 Mar 15. PMID 22422049
- [Background] Green RC, Rehm H, Kohane I. Clinical Genome Sequencing. Genomic and Personalized Medicine 2nd Edition: 102- 122, 2012.
- [Background] Blumenthal-Barby JS, McGuire AL, Green RC, Ubel PA. How behavioral economics can help to avoid 'The last mile problem' in whole genome sequencing. Genome Med. 2015 Jan 22;7(1):3. doi: 10.1186/s13073-015-0132-8. eCollection 2015. PMID 25614766
- [Background] Green RC, Lautenbach D, McGuire AL. GINA, genetic discrimination, and genomic medicine. N Engl J Med. 2015 Jan 29;372(5):397-9. doi: 10.1056/NEJMp1404776. No abstract available. PMID 25629736
- [Result] Vassy JL, Lautenbach DM, McLaughlin HM, Kong SW, Christensen KD, Krier J, Kohane IS, Feuerman LZ, Blumenthal-Barby J, Roberts JS, Lehmann LS, Ho CY, Ubel PA, MacRae CA, Seidman CE, Murray MF, McGuire AL, Rehm HL, Green RC; MedSeq Project. The MedSeq Project: a randomized trial of integrating whole genome sequencing into clinical medicine. Trials. 2014 Mar 20;15:85. doi: 10.1186/1745-6215-15-85. PMID 24645908
- [Result] Vassy JL, McLaughlin HM, MacRae CA, Seidman CE, Lautenbach D, Krier JB, Lane WJ, Kohane IS, Murray MF, McGuire AL, Rehm HL, Green RC. A one-page summary report of genome sequencing for the healthy adult. Public Health Genomics. 2015;18(2):123-9. doi: 10.1159/000370102. Epub 2015 Jan 21. PMID 25612602
- [Derived] Cirino AL, Lakdawala NK, McDonough B, Conner L, Adler D, Weinfeld M, O'Gara P, Rehm HL, Machini K, Lebo M, Blout C, Green RC, MacRae CA, Seidman CE, Ho CY; MedSeq Project*. A Comparison of Whole Genome Sequencing to Multigene Panel Testing in Hypertrophic Cardiomyopathy Patients. Circ Cardiovasc Genet. 2017 Oct;10(5):e001768. doi: 10.1161/CIRCGENETICS.117.001768. PMID 29030401
- [Derived] Vassy JL, Christensen KD, Schonman EF, Blout CL, Robinson JO, Krier JB, Diamond PM, Lebo M, Machini K, Azzariti DR, Dukhovny D, Bates DW, MacRae CA, Murray MF, Rehm HL, McGuire AL, Green RC; MedSeq Project. The Impact of Whole-Genome Sequencing on the Primary Care and Outcomes of Healthy Adult Patients: A Pilot Randomized Trial. Ann Intern Med. 2017 Jun 27;167(3):159-169. doi: 10.7326/M17-0188. Print 2017 Aug 1. PMID 28654958
- See also: NHGRI — http://www.genome.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant recruitment began in 2012 at Brigham and Women's hospital by letter, email, phone and in person.
Groups:
- Family History + Whole Genome Sequencing: Primary Care: Doctors and their patients receive a Genome Report and an Annotated Family History Report.
  Main Study Experimental: Standard of Care + Whole Genome Sequencing (Genome Report): Doctors and their patients receive a Genome Report and a Family History Report.
  There are two sections of the Genome Report:
  1. The General Genome Report, which includes highly penetrant disease mutations, carrier status for recessive disease, and pharmacogenetic associations.
  2. The Cardiac Risk Supplement, which contains genetic information found in the genome regarding cardiac diseases or a risk of cardiovascular diseases that can help with the care of the patient.
- Family History Only: Primary Care: Doctors and their patients receive an Annotated Family History Report only.
  Active Comparator: Standard of Care Only: Doctors and their patients receive a Family History report only
- Family History + Whole Genome Sequencing: Cardiology: Doctors and their patients receive a Genome Report and an Annotated Family History Report.
  Main Study Experimental: Family History + Whole Genome Sequencing (Genome Report): Doctors and their patients receive a Genome Report and a Family History Report.
  There are two sections of the Genome Report:
  The General Genome Report, which includes highly penetrant disease mutations, carrier status for recessive disease, and pharmacogenetic associations.
  The Cardiac Risk Supplement, which contains genetic information found in the genome regarding cardiac diseases or a risk of cardiovascular diseases that can help with the care of the patient.
  Extension Phase: Experimental: Family History + Whole Genome Sequencing (Genome Report)
  *In the main study participants are randomized between Experimental and Comparator, in the Extension phase of the study all participants are in the Experimental Arm.
- Family History Only: Cardiology: Doctors and their patients receive an Annotated Family History Report only. Active Comparator: Family History Only: Doctors and their patients receive a Family History report only
- Extension Cohort: Family History + Whole Genome Sequencing (Genome Report): Doctors and their African American patients receive a Genome Report and a Family History Report.
  There are two sections of the Genome Report:
  1. The General Genome Report, which includes highly penetrant disease mutations, carrier status for recessive disease, and pharmacogenetic associations.
  2. The Cardiac Risk Supplement, which contains genetic information found in the genome regarding cardiac diseases or a risk of cardiovascular diseases that can help with the care of the patient.
Period: Main Study
Arm/Group | Family History + Whole Genome Sequencing: Primary Care | Family History Only: Primary Care | Family History + Whole Genome Sequencing: Cardiology | Family History Only: Cardiology | Extension Cohort
Started | 51 | 50 | 50 | 52 | 10
Completed | 50 | 50 | 49 | 51 | 6
Not Completed | 1 | 0 | 1 | 1 | 4
Period: Long Term Follow-up
Arm/Group | Family History + Whole Genome Sequencing: Primary Care | Family History Only: Primary Care | Family History + Whole Genome Sequencing: Cardiology | Family History Only: Cardiology | Extension Cohort
Started | 26 | 16 | 25 | 25 | 4
Completed | 26 | 16 | 25 | 25 | 4
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Randomized participants who provided information on the baseline survey (main study), or participants who attended disclosure sessions (extension cohort)
Groups:
- Family History + Whole Genome Sequencing: Primary Care; Family History + Whole Genome Sequencing - Cardiology: Doctors and their patients receive a Genome Report and an Annotated Family History Report.
  Main Study Experimental: Family History + Whole Genome Sequencing (Genome Report): Doctors and their patients receive a Genome Report and a Family History Report.
  There are two sections of the Genome Report:
  1. The General Genome Report, which includes highly penetrant disease mutations, carrier status for recessive disease, and pharmacogenetic associations.
  2. The Cardiac Risk Supplement, which contains genetic information found in the genome regarding cardiac diseases or a risk of cardiovascular diseases that can help with the care of the patient.
  Extension Phase: Experimental: Family History + Whole Genome Sequencing (Genome Report)
  *In the main study participants are randomized between Experimental and Comparator, in the Extension phase of the study all participants are in the Experimental Arm.
- Extension Cohort: Doctors and their patients receive a Genome Report and an Annotated Family History Report.
  There are two sections of the Genome Report:
  1. The General Genome Report, which includes highly penetrant disease mutations, carrier status for recessive disease, and pharmacogenetic associations.
  2. The Cardiac Risk Supplement, which contains genetic information found in the genome regarding cardiac diseases or a risk of cardiovascular diseases that can help with the care of the patient.
     * In the main study, participants are randomized between Experimental and Comparator. For the Extension cohort, all participants receive whole genome sequencing.
- Total: Total of all reporting groups
Arm/Group | Family History + Whole Genome Sequencing: Primary Care | Family History Only: Primary Care | Family History + Whole Genome Sequencing - Cardiology | Family History Only: Cardiology | Extension Cohort | Total
Number analyzed (Participants) | 51 | 50 | 50 | 52 | 10 | 213
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 49 | 47 | 32 | 36 | 10 | 174
  >=65 years | 2 | 3 | 18 | 16 | 0 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.2 (7.0) | 54.6 (7.6) | 55.9 (16.1) | 55.9 (12.2) | 51.4 (8.3) | 55.4 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 30 | 24 | 19 | 7 | 109
  Male | 22 | 20 | 26 | 33 | 3 | 104
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 0 | 1 | 1 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 3 | 0 | 10 | 16
  White | 46 | 43 | 45 | 47 | 0 | 181
  More than one race | 0 | 2 | 0 | 1 | 0 | 3
  Unknown or Not Reported | 1 | 3 | 1 | 3 | 0 | 8
Region of Enrollment [Number; unit: participants]
  United States | 51 | 50 | 50 | 52 | 10 | 213

OUTCOME MEASURES:

1. Primary Outcome: Change in Attitudes and Trust
Description: Adapted measures (Hall, MA, et al. 2006) assessed participants' attitudes toward genetic information, trust of their physicians and the medical system regarding interpretation and use of genetic information. Higher scores on a 12-60 scale represent more positive attitudes and greater trust.
Time Frame: Change at 6-weeks post-results disclosure relative to baseline, administered approx.12.5 months after baseline
Population: Participants who completed the baseline survey and 6 week follow-up survey
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Family History + Whole Genome Sequencing - Cardiology: Doctors and their patients receive a Genome Report and an Annotated Family History Report.
  Main Study Experimental: Family History + Whole Genome Sequencing (Genome Report): Doctors and their patients receive a Genome Report and a Family History Report.
  There are two sections of the Genome Report:
  1. The General Genome Report, which includes highly penetrant disease mutations, carrier status for recessive disease, and pharmacogenetic associations.
  2. The Cardiac Risk Supplement, which contains genetic information found in the genome regarding cardiac diseases or a risk of cardiovascular diseases that can help with the care of the patient.
  Extension Phase: Experimental: Family History + Whole Genome Sequencing (Genome Report)
  *In the main study participants are randomized between Experimental and Comparator Arms, in the Extension phase of the study all participants are in the Experimental Arm.
- Family History Only: Cardiology: Doctors and their patients receive an Annotated Family History Report only.
  Active Comparator: Standard of Care Only: Doctors and their patients receive a Family History report only
Arm/Group | Family History + Whole Genome Sequencing: Primary Care | Family History Only: Primary Care | Family History + Whole Genome Sequencing - Cardiology | Family History Only: Cardiology | Extension Cohort
Number analyzed (Participants) | 50 | 44 | 48 | 46 | 6
units on a scale | 0.0 (5.3) | 0.7 (4.5) | 3.5 (5.1) | 1.8 (3.5) | 1.0 (6.3)

2. Primary Outcome: Change in Self Efficacy
Description: Assessed through a scale developed for the Multiplex Initiative (Kaphingst, K.A., et al. 2012). Higher scores on a 0-24 scale indicate greater confidence in participants' abilities to understand genetic information.
Time Frame: Baseline and 6-months post-results disclosure (6 mos. follow-up administered approx. 17 months after baseline)
Population: Participants randomized to the experimental Family History + Whole Genome Sequencing arm who completed both the baseline and the 6-month follow-up surveys
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Family History + Whole Genome Sequencing: Primary Care; Family History + Whole Genome Sequencing - Cardiology: Doctors and their patients receive a Genome Report and an Annotated Family History Report.
  Main Study Experimental: Family History + Whole Genome Sequencing (Genome Report): Doctors and their patients receive a Genome Report and a Family History Report.
  There are two sections of the Genome Report:
  1. The General Genome Report, which includes highly penetrant disease mutations, carrier status for recessive disease, and pharmacogenetic associations.
  2. The Cardiac Risk Supplement, which contains genetic information found in the genome regarding cardiac diseases or a risk of cardiovascular diseases that can help with the care of the patient.
  Extension Phase: Experimental: Family History + Whole Genome Sequencing (Genome Report)
  *In the main study participants are randomized between Experimental and Comparator Arms, in the Extension phase of the study all participants are in the Experimental Arm.
- Extension Cohort: Standard of Care + Whole Genome Sequencing (Genome Report): Doctors and their African American patients receive a Genome Report and a Family History Report.
  There are two sections of the Genome Report:
  1. The General Genome Report, which includes highly penetrant disease mutations, carrier status for recessive disease, and pharmacogenetic associations.
  2. The Cardiac Risk Supplement, which contains genetic information found in the genome regarding cardiac diseases or a risk of cardiovascular diseases that can help with the care of the patient.
Arm/Group | Family History + Whole Genome Sequencing: Primary Care | Family History + Whole Genome Sequencing - Cardiology | Extension Cohort
Number analyzed (Participants) | 49 | 47 | 7
units on a scale | 0.3 (3.4) | 0.5 (4.3) | 3.1 (5.7)

3. Primary Outcome: Change in Preferences for WGS Information
Description: Through nine novel survey items, participants were asked about their preferences for the types of genetic testing results they would like to receive from their whole genome sequence. Scores on an 0-9 scale represent the change in the number of categories of types of genetic testing results out of 9 that participants wanted to learn about from Baseline to 6-weeks follow-up.
Time Frame: Baseline and 6-weeks post-disclosure (6 wks follow-up administered approx. 12.5 mos. after baseline)
Population: Participants who completed both the baseline and 6-week follow-up surveys
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Family History Only: Primary Care; Family History Only: Cardiology: Doctors and their patients receive an Annotated Family History Report only.
  Active Comparator: Family History Only: Doctors and their patients receive a Family History report only
Arm/Group | Family History + Whole Genome Sequencing: Primary Care | Family History Only: Primary Care | Family History + Whole Genome Sequencing - Cardiology | Family History Only: Cardiology | Extension Cohort
Number analyzed (Participants) | 48 | 42 | 47 | 44 | 6
units on a scale | -.1 (1.5) | 0.2 (2.1) | 0 (2.0) | .4 (2.3) | 0.0 (1.9)

4. Primary Outcome: Change in Perceived Health
Description: A single-item measure assessed how participants perceived their own health on a 1-5 scale. Adapted from the SF-12 (DeSalvo KB, Qual Life Res, 2006). Higher scores indicate more positive perceptions of health at follow-up
Time Frame: Baseline, at the disclosure visit (about 1 hour after results disclosure, avg. 11 mos. after baseline) and 6-months post-disclosure (6 mos. follow-up follow-up administered approx. 17 months after baseline)
Population: Participants who completed the item on patient surveys.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Family History + Whole Genome Sequencing: Primary Care: Doctors and their patients receive a Genome Report and an Annotated Family History Report.
  Main Study Experimental: Family History + Whole Genome Sequencing (Genome Report): Doctors and their patients receive a Genome Report and a Family History Report.
  There are two sections of the Genome Report:
  1. The General Genome Report, which includes highly penetrant disease mutations, carrier status for recessive disease, and pharmacogenetic associations.
  2. The Cardiac Risk Supplement, which contains genetic information found in the genome regarding cardiac diseases or a risk of cardiovascular diseases that can help with the care of the patient.
  Extension Phase: Experimental: Family History + Whole Genome Sequencing (Genome Report)
  *In the main study participants are randomized between Experimental and Active Comparator, in the Extension phase of the study all participants are in the Experimental Arm.
- Family History + Whole Genome Sequencing: Cardiology: Doctors and their patients receive a Genome Report and an Annotated Family History Report.
  Main Study Experimental: Family History + Whole Genome Sequencing (Genome Report): Doctors and their patients receive a Genome Report and a Family History Report.
  There are two sections of the Genome Report:
  1. The General Genome Report, which includes highly penetrant disease mutations, carrier status for recessive disease, and pharmacogenetic associations.
  2. The Cardiac Risk Supplement, which contains genetic information found in the genome regarding cardiac diseases or a risk of cardiovascular diseases that can help with the care of the patient.
  Extension Phase: Experimental: Family History + Whole Genome Sequencing (Genome Report)
  *In the main study participants are randomized between Experimental and Active Comparator arms, in the Extension phase of the study all participants are in the Experimental Arm.
Arm/Group | Family History + Whole Genome Sequencing: Primary Care | Family History Only: Primary Care | Family History + Whole Genome Sequencing: Cardiology | Family History Only: Cardiology | Extension Cohort
Number analyzed (Participants) | 50 | 49 | 49 | 51 | 8
units on a scale
  Change at disclosure | -0.1 (0.6) | 0 (0.6) | 0 (0.6) | -0.2 (0.7) | 0.3 (0.5)
  Change at 6 months post-disclosure: number analyzed (Participants) | 49 | 44 | 47 | 49 | 7
  Change at 6 months post-disclosure | -0.1 (0.7) | -0.1 (0.7) | -0.1 (0.8) | -0.3 (0.8) | 0.1 (0.4)

5. Primary Outcome: Change in Shared Decision Making
Description: Changes in shared decision making were assessed through a single item adapted from the Control Preferences Scale, a measure designed to ascertain the degree of control an individual wants to assume when decisions are being made about medical treatment. Higher scores on a scale of 1-3 indicate preferences towards more equally shared decision making (Heisler et al 2003). Higher mean changes over time indicate a change in preference towards more equally shared decision making at follow-up.
Time Frame: Baseline and 6-weeks post-disclosure (6 wks follow-up administered approx. 12.5 mos. after baseline)
Population: Participants who were completed the item on both the baseline and 6-week follow-up surveys
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Family History Only: Cardiology: Doctors and their patients receive an Annotated Family History Report only.
  Placebo Comparator: Family History Only: Doctors and their patients receive a Family History report only
Arm/Group | Family History + Whole Genome Sequencing: Primary Care | Family History Only: Primary Care | Family History + Whole Genome Sequencing - Cardiology | Family History Only: Cardiology | Extension Cohort
Number analyzed (Participants) | 46 | 41 | 46 | 45 | 5
units on a scale | 0.1 (0.7) | 0 (0.5) | 0.2 (0.8) | 0.1 (0.7) | -0.2 (0.8)

6. Primary Outcome: Change in Intolerance of Uncertainty
Description: Changes in participants' tolerance for uncertainty were assessed through a short 12-item version of the Intolerance of Uncertainty Scale (Carleton, 2007). Total summed scale range is 12-60, with higher scores indicating increased negative feelings about uncertainty from baseline to follow-up.
Time Frame: Baseline and 6-months post-disclosure (6 mos. follow-up administered approx. 17 mos. after baseline)
Population: Participants who completed both the baseline and 6-month follow-up surveys
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History + Whole Genome Sequencing: Primary Care | Family History Only: Primary Care | Family History + Whole Genome Sequencing - Cardiology | Family History Only: Cardiology | Extension Cohort
Number analyzed (Participants) | 49 | 44 | 47 | 49 | 7
units on a scale | -0.5 (6.3) | 0.3 (6.6) | -1.3 (5.8) | 0 (7.4) | 4.9 (14.4)

7. Primary Outcome: Change in General Anxiety and Depression
Description: The Hospital Anxiety and Depression Scale (HADS) scale was administered through a survey. This is a validated scale designed to assess the participants' level of depression and anxiety through Likert-type questions. Total ranges for each summed subscale, anxiety and depression, is 0-21. Any participant scoring >14 on the anxiety subscale or >16 on the depression subscale were contacted by study staff for evaluation. Higher scores indicate increased anxiety or depression from baseline to follow-up.
Time Frame: Baseline, at the disclosure visit (about 1 hour after results disclosure, avg. 11 mos. after baseline), 6-weeks post-disclosure and 6-months post-disclosure (6 wks. follow-up administered approx. 12.5 mos and 6 mos follow-up approx 17 mos. after baseline)
Population: Participants who completed the baseline survey and follow-up surveys
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History + Whole Genome Sequencing: Primary Care | Family History Only: Primary Care | Family History + Whole Genome Sequencing - Cardiology | Family History Only: Cardiology | Extension Cohort
Number analyzed (Participants) | 50 | 49 | 49 | 51 | 8
units on a scale
  Change in Anxiety at disclosure | 0.1 (2.3) | -.2 (2.8) | -.4 (1.9) | -.3 (2.8) | -0.5 (1.5)
  Change in Anxiety at 6 Weeks: number analyzed (Participants) | 50 | 44 | 48 | 46 | 6
  Change in Anxiety at 6 Weeks | -1.4 (3.2) | -.8 (2.3) | -1.7 (2.6) | -1.0 (2.4) | -1.5 (1.5)
  Change in Anxiety at 6 Months: number analyzed (Participants) | 49 | 44 | 47 | 49 | 7
  Change in Anxiety at 6 Months | -.2 (2.6) | -.1 (2.6) | -.2 (2.4) | -.4 (2.4) | -0.9 (3.0)
  Change in Depression at disclosure | 0 (2.1) | 0.7 (2.6) | -0.1 (1.6) | 0 (2.0) | -0.3 (2.8)
  Change in Depression at 6 Weeks: number analyzed (Participants) | 50 | 44 | 48 | 46 | 6
  Change in Depression at 6 Weeks | -.3 (2.1) | 0.4 (2.7) | -.8 (1.7) | -.2 (1.8) | -1.0 (2.8)
  Change in Depression at 6 Months: number analyzed (Participants) | 49 | 44 | 47 | 49 | 7
  Change in Depression at 6 Months | -.1 (1.9) | 0.5 (2.1) | -.1 (1.9) | 0 (1.8) | 0.9 (3.8)

8. Primary Outcome: Change in Health Behaviors
Description: Novel items that asked whether participants changed vitamin use, supplement use, medication use, diet, exercise, or "other" health behaviors. Counts and percentages represent participants who reported any health behavior changes.
Time Frame: 6-weeks post-disclosure and 6-months post-disclosure (6 wks. follow-up administered approx. 12.5 mos. and 6 mos. follow-up approx. 17 mos. after baseline)
Population: Participants who attended disclosure sessions and responded to post-disclosure surveys
Measure: Count of Participants; unit: Participants
Arm/Group | Family History + Whole Genome Sequencing: Primary Care | Family History Only: Primary Care | Family History + Whole Genome Sequencing - Cardiology | Family History Only: Cardiology | Extension Cohort
Number analyzed (Participants) | 50 | 44 | 48 | 49 | 7
Participants
  6 Weeks Post-Disclosure: number analyzed (Participants) | 50 | 43 | 48 | 46 | 6
  6 Weeks Post-Disclosure | 24 | 16 | 17 | 15 | 4
  6 Months Post-Disclosure: number analyzed (Participants) | 49 | 44 | 47 | 49 | 7
  6 Months Post-Disclosure | 20 | 13 | 26 | 20 | 3

9. Primary Outcome: Information Sharing
Description: Sharing of information was assessed by asking patients if they intended to share results with others (at the end of the disclosure visit) and if they had shared their results with others (6 months after disclosure) adapted from the Health Information National Trends Survey (HINTS).
Time Frame: At the disclosure visit (about 1 hour after results disclosure, avg. 11 mos. after baseline) and 6-months post-disclosure (approx. 17 mos. after baseline)
Population: Participants who answered information-sharing questions on the post-disclosure or 6-month follow-up questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Family History + Whole Genome Sequencing: Primary Care | Family History Only: Primary Care | Family History + Whole Genome Sequencing - Cardiology | Family History Only: Cardiology | Extension Cohort
Number analyzed (Participants) | 46 | 47 | 43 | 45 | 7
Participants
  Plans to share at disclosure: number analyzed (Participants) | 44 | 47 | 43 | 41 | 7
  Plans to share at disclosure | 43 | 39 | 42 | 30 | 6
  Shared, per 6 month survey: number analyzed (Participants) | 46 | 39 | 39 | 45 | 5
  Shared, per 6 month survey | 41 | 27 | 38 | 28 | 4

10. Primary Outcome: Changes in Genomic Literacy
Description: Changes in participants' genomic literacy were measured with an 11-item measure adapted from the ClinSeq Study (Kaphingst K.A. et al. 2012) administered at baseline and 6 months post-disclosure. Items are marked as correct (1) or incorrect (0) and summed for a total scale range of 0 to 11, with higher scores indicating higher genomic literacy.
Time Frame: Assessing Genomic Literacy at baseline and 6-months post-disclosure (approx. 17 mos. after baseline)
Population: Participants who completed the genetic literacy items in the baseline and 6-month follow-up surveys
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History + Whole Genome Sequencing: Primary Care | Family History Only: Primary Care | Family History + Whole Genome Sequencing - Cardiology | Family History Only: Cardiology | Extension Cohort
Number analyzed (Participants) | 50 | 45 | 47 | 49 | 7
units on a scale | -.4 (1.8) | -.5 (2.3) | -.6 (2.1) | -.2 (1.2) | 0.0 (1.6)

11. Primary Outcome: Changes in Health Care Utilization
Description: Participants' health care utilization was assessed through a combination of medical record reviews and novel and adapted measures from the Behavioral Risk Factor Surveillance System (BRFSS). Changes are assessed by comparing the number of services and procedures received in 6 months following disclosure against the number of services and procedures received in the 6 months prior to disclosure.
Time Frame: 6 months prior to disclosure and 6-months post-disclosure (approx. 17 mos. after baseline) and 5-years post-disclosure
Population: All randomized participants who received disclosure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History + Whole Genome Sequencing: Primary Care | Family History Only: Primary Care | Family History + Whole Genome Sequencing - Cardiology | Family History Only: Cardiology | Extension Cohort
Number analyzed (Participants) | 50 | 50 | 49 | 51 | 10
units on a scale
  Visits | 3.9 (7.9) | 2.3 (6.8) | 1.7 (7.8) | 1.7 (7.1) | 0.6 (3.7)
  Labs: number analyzed (Participants) | 50 | 50 | 49 | 51 | 5
  Labs | 1.4 (8.9) | -0.3 (7.8) | 1.5 (10.6) | 1.5 (7.4) | 0.5 (1.2)
  Imaging tests | 0 (2.1) | -.1 (2.6) | 0.9 (2.1) | 1.0 (1.7) | 0.0 (0.0)
  Cardiology tests: number analyzed (Participants) | 50 | 50 | 49 | 51 | 6
  Cardiology tests | 0.2 (1.0) | 0.2 (0.8) | 0.8 (2.7) | 0.9 (3.0) | 0.3 (0.6)
  Hospitalizations | 0 (0.1) | 0 (0.2) | 0.1 (0.6) | 0.1 (0.7) | 0.0 (0.0)

12. Primary Outcome: Change in Perceived Utility
Description: A novel survey item asked participants to rate the usefulness of whole genome sequencing results for managing health on a 1-10 scale. Scores at 6 months were compared to scores at baseline.
Time Frame: At baseline and 6-months post-disclosure (approx. 17 mos. after baseline)
Population: Participants who received whole genome sequencing and completed the survey items at baseline and at 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History + Whole Genome Sequencing: Primary Care | Family History + Whole Genome Sequencing - Cardiology | Extension Cohort
Number analyzed (Participants) | 48 | 45 | 7
units on a scale | -.6 (2.5) | -.9 (3.0) | -1.0 (2.3)

13. Secondary Outcome: Psychological Impact
Description: Psychological impact was assessed by a modified version of the Multidimensional Impact of Cancer Risk Assessment (MICRA) questionnaire. Higher scores indicated more distress related to study results.
Time Frame: 6-weeks post-disclosure and 6-months post-disclosure (6wks. follow-up administered approx. 12.5 mos. and 6 mos. follow-up approx. 17 mos. after baseline)
Population: Participants who answered the psychological impact items on the 6 week or 6 month follow-up questionnaires
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History + Whole Genome Sequencing: Primary Care | Family History Only: Primary Care | Family History + Whole Genome Sequencing - Cardiology | Family History Only: Cardiology | Extension Cohort
Number analyzed (Participants) | 46 | 41 | 45 | 44 | 7
units on a scale
  6 Weeks Post-Disclosure: number analyzed (Participants) | 46 | 37 | 45 | 43 | 6
  6 Weeks Post-Disclosure | 13.2 (3.8) | 15.1 (3.9) | 14.2 (4.8) | 14.5 (4.3) | 11.4 (4.2)
  6 Months Post-Disclosure: number analyzed (Participants) | 42 | 41 | 45 | 44 | 7
  6 Months Post-Disclosure | 14.9 (3.2) | 15.2 (3.7) | 16.0 (5.4) | 16.5 (5.6) | 14.1 (3.5)

14. Secondary Outcome: Decisional Regret
Description: Participants' satisfaction with their decision to participate in the MedSeq Project through a 5-item validated scale (Brehaut 2003). Average score computed after reversing scores of 2 negatively phrased items and converting score to range from 0-100 by subtracting 1 and multiplying by 25. Higher scores indicate greater regret.
Time Frame: At post-disclosure visit (about 1 hour after results disclosure, avg. 11 mos. after baseline), at 6-weeks post-disclosure, and at 6-months post-disclosure (6 wks follow-up approx. 12.5 mos. and 6 mos. follow-up approx. 17 mos. after baseline)
Population: Participants who answered the decisional regret items on the post-disclosure, 6 week follow-up, or 6 month follow-up surveys
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History + Whole Genome Sequencing: Primary Care | Family History Only: Primary Care | Family History + Whole Genome Sequencing - Cardiology | Family History Only: Cardiology | Extension Cohort
Number analyzed (Participants) | 50 | 49 | 49 | 51 | 9
units on a scale
  Post-Disclosure | 8.9 (16.7) | 12.9 (14.0) | 6.2 (9.6) | 15.8 (22.8) | 6.1 (10.8)
  6 Weeks Post-Disclosure: number analyzed (Participants) | 50 | 44 | 48 | 46 | 7
  6 Weeks Post-Disclosure | 9.8 (16.6) | 17.2 (15.5) | 5.8 (9.7) | 15.0 (20.6) | 6.4 (11.1)
  6 Months Post-Disclosure: number analyzed (Participants) | 50 | 45 | 47 | 49 | 6
  6 Months Post-Disclosure | 11.5 (18.2) | 19.9 (19.3) | 7.9 (11.2) | 11.3 (15.9) | 4.2 (10.2)

15. Secondary Outcome: Understanding
Description: A novel item assessed participants' subjective understanding of their study results on a 1-5 scale, where higher scores indicate greater subjective understanding.
Time Frame: as for outcome 14
Population: Participants who answered the understanding item on the post-disclosure, 6-week follow-up, or 6-month follow-up surveys.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History + Whole Genome Sequencing: Primary Care | Family History Only: Primary Care | Family History + Whole Genome Sequencing - Cardiology | Family History Only: Cardiology | Extension Cohort
Number analyzed (Participants) | 50 | 44 | 49 | 49 | 7
units on a scale
  Post-Disclosure: number analyzed (Participants) | 49 | 32 | 49 | 35 | 7
  Post-Disclosure | 4.2 (0.7) | 4.5 (0.7) | 4.0 (0.7) | 4.2 (0.8) | 3.9 (0.7)
  6 Weeks Post-Disclosure: number analyzed (Participants) | 50 | 43 | 48 | 46 | 7
  6 Weeks Post-Disclosure | 4.2 (0.8) | 4.2 (0.9) | 4.1 (0.7) | 4.2 (0.9) | 4.0 (0.6)
  6 Months Post-Disclosure: number analyzed (Participants) | 50 | 44 | 47 | 49 | 7
  6 Months Post-Disclosure | 4.0 (0.7) | 4.3 (0.7) | 4.0 (0.8) | 4.2 (0.7) | 4.0 (0.6)

16. Secondary Outcome: Expectations
Description: Novel survey items asked participants about whether or not their genetic test results would be useful for specific reasons. Response options were "no," "probably not", "probably yes," and "yes." Responses of "probably yes" and "yes" were combined to simplify presentation of data.
Time Frame: Baseline
Population: Randomized participants who completed the baseline survey.
Measure: Count of Participants; unit: Participants
Groups:
- Family History + Whole Genome Sequencing - Cardiology: Doctors and their patients receive a Genome Report and an Annotated Family History Report.
  Main Study Experimental: Family History + Whole Genome Sequencing (Genome Report): Doctors and their patients receive a Genome Report and a Family History Report.
  There are two sections of the Genome Report:
  1. The General Genome Report, which includes highly penetrant disease mutations, carrier status for recessive disease, and pharmacogenetic associations.
  2. The Cardiac Risk Supplement, which containd genetic information found in the genome regarding cardiac diseases or a risk of cardiovascular diseases that can help with the care of the patient.
  Extension Phase: Experimental: Family History + Whole Genome Sequencing (Genome Report)
  *In the main study participants are randomized between Experimental and Comparator arms, in the Extension phase of the study all participants are in the Experimental Arm.
Arm/Group | Family History + Whole Genome Sequencing: Primary Care | Family History Only: Primary Care | Family History + Whole Genome Sequencing - Cardiology | Family History Only: Cardiology | Extension Cohort
Number analyzed (Participants) | 51 | 49 | 50 | 52 | 10
Participants
  Identify disease risk: number analyzed (Participants) | 51 | 48 | 48 | 52 | 10
  Identify disease risk | 40 | 36 | 41 | 42 | 8
  Influence treatment | 43 | 44 | 41 | 44 | 10
  Influence medical care: number analyzed (Participants) | 51 | 49 | 48 | 52 | 10
  Influence medical care | 44 | 46 | 40 | 44 | 9
  Influence medications: number analyzed (Participants) | 50 | 49 | 50 | 52 | 10
  Influence medications | 35 | 41 | 36 | 35 | 10
  Influence end-of-life planning: number analyzed (Participants) | 51 | 49 | 49 | 52 | 10
  Influence end-of-life planning | 27 | 19 | 25 | 22 | 7
  Influence reproductive decisions: number analyzed (Participants) | 51 | 48 | 50 | 52 | 10
  Influence reproductive decisions | 18 | 8 | 24 | 16 | 4

ADVERSE EVENTS:
Time Frame: Baseline to 6 months for the main cohort and through 5 years for the Long Term Follow-up cohort
Description: Adverse event definitions are consistant with clinicatrials.gov
  Adverse events were collected and reported to the IRB
Groups:
- Family History + Whole Genome Sequencing: Cardiology: Doctors and their patients receive a Genome Report and an Annotated Family History Report.
  Main Study Experimental: Family History + Whole Genome Sequencing (Genome Report): Doctors and their patients receive a Genome Report and a Family History Report.
  There are two sections of the Genome Report:
  1. The General Genome Report, which includes highly penetrant disease mutations, carrier status for recessive disease, and pharmacogenetic associations.
  2. The Cardiac Risk Supplement, which contains genetic information found in the genome regarding cardiac diseases or a risk of cardiovascular diseases that can help with the care of the patient.
  Extension Phase: Experimental: Family History + Whole Genome Sequencing (Genome Report)
  *In the main study participants are randomized between Experimental and Comparator arms, in the Extension phase of the study all participants are in the Experimental Arm.
- Extension Cohort: Family History + Whole Genome Sequencing (Genome Report): Doctors and their African American patients receive a Genome Report and a Family History Report.
  There are two sections of the Genome Report:
  The General Genome Report, which includes highly penetrant disease mutations, carrier status for recessive disease, and pharmacogenetic associations.
  The Cardiac Risk Supplement, which contains genetic information found in the genome regarding cardiac diseases or a risk of cardiovascular diseases that can help with the care of the patient.
Arm/Group | Family History + Whole Genome Sequencing: Primary Care | Family History Only: Primary Care | Family History + Whole Genome Sequencing: Cardiology | Family History Only: Cardiology | Extension Cohort
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/50 | 3/50 | 1/52 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/50 | 3/50 | 1/52 | 0/10
Other Adverse Events (participants affected / at risk) | 0/51 | 3/50 | 0/50 | 0/52 | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Family History + Whole Genome Sequencing: Primary Care (N=51) | Family History Only: Primary Care (N=50) | Family History + Whole Genome Sequencing: Cardiology (N=50) | Family History Only: Cardiology (N=52) | Extension Cohort (N=10)
Serious (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) — Deceased- Complications of Cardiomyopathy
Death (Cardiac disorders) | NA | NA | 3 | 1 | NA — Learned that participant had died when called to collect long term follow-up data. Cause of death from medical record review appears to be a stroke. Not related to the intervention
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Family History + Whole Genome Sequencing: Primary Care (N=51) | Family History Only: Primary Care (N=50) | Family History + Whole Genome Sequencing: Cardiology (N=50) | Family History Only: Cardiology (N=52) | Extension Cohort (N=10)
Other (Psychiatric disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) — Elevated HADS scale anxiety score

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-25): https://cdn.clinicaltrials.gov/large-docs/66/NCT01736566/Prot_SAP_000.pdf